CLINICAL TRIAL: NCT05531305
Title: Longitudinal Changes in Muscle Mass After Intensive Care: a Pilot Feasibility Study.
Brief Title: Longitudinal Changes in Muscle Mass After Intensive Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Martin Sundstrom Rehal, Principal Investigator, Karolinska University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: K 2022-6873
Record Dates: First submitted 2022-09-02; First posted 2022-09-07 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Critical Illness; Muscle Loss
MeSH Terms: conditions — Critical Illness; Muscular Atrophy | interventions — Calorimetry, Indirect

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study intervention (Experimental)
  Interventions: Device: Muscle ultrasound; Device: Indirect calorimetry; Diagnostic Test: Hand dynamometry; Diagnostic Test: MRC Sum Score

INTERVENTIONS:
Device: Muscle ultrasound — Standardized ultrasonographic measurement of quadriceps muscle layer thickness.
Device: Indirect calorimetry — Non-invasive measurement of resting energy expenditure using the Q-NRG metabolic monitor with hood and canopy.
Diagnostic Test: Hand dynamometry — Assessment of handgrip strength using hand dynamometry.
Diagnostic Test: MRC Sum Score — Assessment of muscle function/limb strength using the Medical Research Council sum score (12-60 points).

SUMMARY:
Critically ill patients often suffer from dramatic muscle loss while in the ICU. Recovery of muscle structure and function have been proposed as core outcome measures for interventional studies in ICU survivors. Ultrasound is an accessible and validated tool to monitor muscle mass over time, with quadriceps muscle layer thickness (MLT) corresponding well to more invasive or cumbersome modalities. In order to design adequately powered studies investigating the effects of nutritional or metabolic interventions on post-ICU recovery, an estimate of the population standard deviation in MLT change over time is required. Currently there is a paucity of data describing changes in muscle mass during the subsequent period of hospitalization in ICU survivors.

The aim of this study is to estimate the mean change and standard deviation in quadriceps MLT over time, in patients discharged alive from intensive care. Patients will be followed until hospital discharge or up to 28 days after ICU discharge. Interactions with nutritional intake, inflammation and metabolic rate will be analyzed for hypothesis-generating purposes.

DETAILED DESCRIPTION:
Background

Rapid and severe muscle loss is a common feature in intensive care [1]. Nutritional support is provided with the intention of preventing excessive muscle protein breakdown, but the evidence that higher energy or protein intake can mitigate muscle wasting in the ICU is limited [2]. A potential explanation to these findings is the proinflammatory and catabolic state often associated with critical illness [3]. As long as a patient remains critically ill, the potential to promote anabolism and recovery may be limited.

It is well-documented that patients discharged from ICU often suffer from poor oral intake during hospital stay [4,5]. Optimizing nutritional support in the post-ICU period may therefore be a simple and cost-effective way of counteracting sarcopenia and improving health-related outcomes [6]. Currently there is a lack of published studies investigating the effect of nutritional interventions on lean body mass after intensive care. This may be due to the cumbersome and resource-intensive methods previously available for measuring body composition. In recent years, bedside ultrasound has become increasingly popular as a research tool for monitoring muscle loss over time. It has been validated against other radiological modalities, is non-invasive and accessible [7].

As there is a lack of literature describing sonographic changes in muscle mass over time in the post-ICU phase, data is needed to support a formal power calculation for interventional studies assessing muscle loss as a primary outcome measure. We therefore plan an observational longitudinal study to describe the change in quadriceps muscle layer thickness over time between ICU and hospital discharge.

Aim

The aims of this project are to 1) estimate the standard deviation of the change in quadriceps muscle layer thickness (MLT) over time, and 2) determine the feasibility of performing a longitudinal follow-up of MLT and energy expenditure in hospitalized patients after ICU discharge.

Hypothesis

In patients discharged alive from the ICU, there is a decrease in mean MLT over time during hospitalization

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old.
* ICU length of stay ≥3 days.
* Expected to be discharged alive within 72 hours.

Exclusion Criteria:

* Lack of informed consent.
* Limitations in treatment to best supportive care (not expected to survive hospitalization).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

PRIMARY OUTCOMES:
Quadriceps muscle layer thickness (MLT) | From ICU discharge to either hospital discharge or up to 28 days after ICU discharge, whichever comes first. The first measurement is performed within 72 hours after ICU discharge and repeated every 3-5 days.
  Change in quadriceps MLT (mean +/- standard deviation) over time.

SECONDARY OUTCOMES:
Resting energy expenditure (REE) | From ICU discharge to either hospital discharge or up to 28 days after ICU discharge, whichever comes first. The first measurement is performed within 72 hours after ICU discharge and repeated every 3-5 days.
  Change in REE over time.

OTHER OUTCOMES:
Handgrip strength | From ICU discharge to either hospital discharge or up to 28 days after ICU discharge, whichever comes first. The first measurement is performed within 72 hours after ICU discharge and repeated every 3-5 days.
  Change in handgrip strength, as assessed by hand dynamometry, over time.
MRC sum score | From ICU discharge to either hospital discharge or up to 28 days after ICU discharge, whichever comes first. The first assessment is performed within 72 hours after ICU discharge and repeated every 3-5 days.
  Change in MRC sum score over time.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Sundström Rehal, MD PhD, Principal Investigator — Karolinska University Hospital; Olav Rooyackers, PhD, Study Chair — Karolinska Institutet
Locations (1):
- Karolinska University Hospital, Huddinge, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies TW, van Gassel RJJ, van de Poll M, Gunst J, Casaer MP, Christopher KB, Preiser JC, Hill A, Gundogan K, Reintam-Blaser A, Rousseau AF, Hodgson C, Needham DM, Castro M, Schaller S, McClelland T, Pilkington JJ, Sevin CM, Wischmeyer PE, Lee ZY, Govil D, Li A, Chapple L, Denehy L, Montejo-Gonzalez JC, Taylor B, Bear DE, Pearse R, McNelly A, Prowle J, Puthucheary ZA. Core outcome measures for clinical effectiveness trials of nutritional and metabolic interventions in critical illness: an international modified Delphi consensus study evaluation (CONCISE). Crit Care. 2022 Aug 6;26(1):240. doi: 10.1186/s13054-022-04113-x. PMID 35933433
- [Background] Puthucheary ZA, Rawal J, McPhail M, Connolly B, Ratnayake G, Chan P, Hopkinson NS, Phadke R, Dew T, Sidhu PS, Velloso C, Seymour J, Agley CC, Selby A, Limb M, Edwards LM, Smith K, Rowlerson A, Rennie MJ, Moxham J, Harridge SD, Hart N, Montgomery HE. Acute skeletal muscle wasting in critical illness. JAMA. 2013 Oct 16;310(15):1591-600. doi: 10.1001/jama.2013.278481. PMID 24108501
- [Background] Preiser JC, Ichai C, Orban JC, Groeneveld AB. Metabolic response to the stress of critical illness. Br J Anaesth. 2014 Dec;113(6):945-54. doi: 10.1093/bja/aeu187. Epub 2014 Jun 26. PMID 24970271
- [Background] Fischer A, Hertwig A, Hahn R, Anwar M, Siebenrock T, Pesta M, Liebau K, Timmermann I, Brugger J, Posch M, Ringl H, Tamandl D, Hiesmayr M; USVALID Collaboration Group. Validation of bedside ultrasound to predict lumbar muscle area in the computed tomography in 200 non-critically ill patients: The USVALID prospective study. Clin Nutr. 2022 Apr;41(4):829-837. doi: 10.1016/j.clnu.2022.01.034. Epub 2022 Feb 11. PMID 35263692
- [Background] Ridley EJ, Parke RL, Davies AR, Bailey M, Hodgson C, Deane AM, McGuinness S, Cooper DJ. What Happens to Nutrition Intake in the Post-Intensive Care Unit Hospitalization Period? An Observational Cohort Study in Critically Ill Adults. JPEN J Parenter Enteral Nutr. 2019 Jan;43(1):88-95. doi: 10.1002/jpen.1196. Epub 2018 Jun 20. PMID 29924393
- [Background] Schuetz P, Fehr R, Baechli V, Geiser M, Deiss M, Gomes F, Kutz A, Tribolet P, Bregenzer T, Braun N, Hoess C, Pavlicek V, Schmid S, Bilz S, Sigrist S, Brandle M, Benz C, Henzen C, Mattmann S, Thomann R, Brand C, Rutishauser J, Aujesky D, Rodondi N, Donze J, Stanga Z, Mueller B. Individualised nutritional support in medical inpatients at nutritional risk: a randomised clinical trial. Lancet. 2019 Jun 8;393(10188):2312-2321. doi: 10.1016/S0140-6736(18)32776-4. Epub 2019 Apr 25. PMID 31030981
- [Derived] Sundstrom Rehal M, Sebghati Sparrfelt C, Lajewska N, Fischer A, Kilsand K, Helleberg J, Habel H, Rooyackers O. Longitudinal changes in muscle mass after ICU discharge: A prospective observational cohort study. Clin Nutr. 2025 Nov;54:53-61. doi: 10.1016/j.clnu.2025.09.004. Epub 2025 Sep 18. PMID 41027230